CLINICAL TRIAL: NCT01111877
Title: Natural History Study of Incidence of Otorrhea Following Tympanostomy Tube Insertion in Children 6 Months to 12 Years
Status: Terminated | Type: Observational
Why Stopped: Management Decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: C-09-041
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Otorrhea
Keywords: ear tubes; ear drainage; ear infection; ear drops; tympanostomy tubes; Pediatric patients
MeSH Terms: conditions — Otitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
This study was conducted to describe the time to first incidence of otorrhea post tympanostomy tube insertion.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 6 months old and no more than 13 years of age at the time of enrollment scheduled for unilateral or bilateral myringotomy and tympanostomy tube insertion. Patients and/or child must read/sign informed consent and comply with requirement of the study.

Exclusion Criteria:

* There are no exclusion criteria.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients between the ages of 6 months and 12 years who are undergoing unilateral or bilateral myringotomy with placement of tympanostomy tube.
Sampling Method: Non-Probability Sample
Enrollment: 1389 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Incidence of, time to, and relationship of risk factors associated with otorrhea post tympanostomy tube insertion. | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States